CLINICAL TRIAL: NCT03320356
Title: Transcultural Validation of the Oxford Shoulder Score for the French-speaking Population
Acronym: French-OSS
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2016Ao001
Record Dates: First submitted 2017-10-17; First posted 2017-10-25 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- shoulder pain: Patients presenting inflammatory, degenerative, or post-traumatic shoulder pain and consulting at Orthopaedic Department, Reims Teaching Hospital.
  Interventions: Other: the French version of the Oxford Shoulder Score

INTERVENTIONS:
Other: the French version of the Oxford Shoulder Score

SUMMARY:
Degenerative lesions of the shoulder occur very frequently and their incidence increases with age. The Constant-Murley score is currently considered the gold standard in Europe to assess the shoulder and is widely used by the orthopaedic community to follow up on shoulder pathologies. However, healthcare professionals are taking an increasing interest in self-administered patient-reported out-come measures. Several self-administered questionnaires are available to assess the shoulder. Among these questionnaires, the OSS (Oxford Shoulder Score) is considered to be quick, simple, and reliable for the English-speaking population. This score was initially developed at the University of Oxford in 1996. It is a self-administered questionnaire designed to evaluate pain and shoulder function through 12 questions. This score has since been adapted in different languages but not in French.

DETAILED DESCRIPTION:
The aim was to develop a translation and a transcultural adaptation of the OSS and to assess its validity in native French-speaker patients with shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving chemotherapy for solid tumors in Ambulatory Medicine Unit of the Reims University Hospital (France) between May 14, 2012 and July 31, 2013
* native French speakers

Exclusion Criteria:

* Patients who presented shoulder's instability problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting inflammatory, degenerative, or post-traumatic shoulder pain and consulting at Orthopaedic Department, Reims Teaching Hospital (France) between November, 2014 and March, 2015.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Acceptability of the French version of the Oxford Shoulder Score | Day 0
  Acceptability was analysed using the rate of refusal to participate. It is a 12-item self-administered questionnaire developed for patients with inflammatory or degenerative shoulder disease.
  Each question presents five possible responses corresponding to a score of 0 (worst situation) to 4 (best situation). Questionnaire produces a single score with a range from 0 (least difficulties) to 48 (most difficulties).
Feasibility of the French version of the Oxford Shoulder Score | Day 0
  Feasibility was analysed using the nonresponse rate. It is a 12-item self-administered questionnaire developed for patients with inflammatory or degenerative shoulder disease.
  Each question presents five possible responses corresponding to a score of 0 (worst situation) to 4 (best situation). Questionnaire produces a single score with a range from 0 (least difficulties) to 48 (most difficulties).

SECONDARY OUTCOMES:
Convergent validity of the French version of the Oxford Shoulder Score | Day 0
  The convergent validity was studied using correlation between the Oxford Shoulder Score and the Constant score and between the Oxford Shoulder Score and the Subjective Shoulder Score score.
test/retest reliability of the French version of the Oxford Shoulder Score | Day 0
  Test/retest reliability was analysed using calculation of the intraclass correlation coefficient. An ICC > 0.8 indicates good test/retest reliability.
Internal coherence of the French version of the Oxford Shoulder Score | Day 0
  The internal coherence was tested using the Cronbach coefficient. The acceptable threshold for internal coherence was a Cronbach coefficient equal or more than 0.7

REFERENCES:
- [Result] Tuton D, Barbe C, Salmon JH, Drame M, Nerot C, Ohl X. Transcultural validation of the Oxford Shoulder Score for the French-speaking population. Orthop Traumatol Surg Res. 2016 Sep;102(5):555-8. doi: 10.1016/j.otsr.2016.05.010. Epub 2016 Jul 22. PMID 27460650